CLINICAL TRIAL: NCT03976661
Title: Measuring the Impact of Taking Care in the Context of an Innovative System for Keeping Dependent Elderly People in Their Homes
Acronym: DIAPASON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A03183-52
Record Dates: First submitted 2019-06-04; First posted 2019-06-06 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Patient With no Severe Behavioural Disorders and Whose Situation Would Require Entry Into Classique EHPAD (Retirement Home)
Keywords: No severe behavioural disorders, EHPAD (retirement home), Older patients, loss of autonomy, Groupe-Iso-Ressources (GIR)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DIAPASON 92 arm: Arm will be constitued by older patients with loss of autonomy, living at home benefiting from the device DIAPASON 92 (Innovative support system for elderly people in their homes)
- Control arm: Arm will be constituted by people residing at the EHPAD (retirement home)

SUMMARY:
The purpose of this study is to compare life quality of patients taking care by DIAPASON 92 with patients or residents from control group EHPAD (retirement home)

DETAILED DESCRIPTION:
This study has two components: a quantitative component(for users and caregivers) and a qualitative component (for users, caregivers and professionals)

About population :

For quantitative component: the investigators have two arms:

* Diapason 92 arm: will be constitued by older patients with loss of autonomy, living at home and benefiting from Diapason 92 device
* Control arm: will be constituted by people residing at the EHPAD (retirement home)

For qualitative component: Study will cover 5 different populations since it concerns both:- - Diapason 92 professionals who work directly with users

* Daipason 92 Supervisory staff
* Diapason 92 professional partners, including referring physicians.
* The users
* Non-professional helpers of users

Conduct of study:

- About quantitative component:

After verification of eligibility criteria adapted to each centre and once the non-opposition has been collected and subjects have been included, the following data will be collected at M0, M3, M6 and M12:

* For patients : Start date of care by Diapason 92 or EHPAD, Quality of Life score, benefit evaluation, Socio-educational level, evaluation of disruptive behaviour disorders, economic indicators, somatic comorbidities, collection of psychiatric follow-up if available, independence, nutritional status, factors(s) that motivated care, cognitive assessment, balance assessment, depression screening, ergonomic assessment (only for Diapason 92
* Family caregiver: 3 measures will be collected: Measuring the burden by Zarit scale, self-assessment of his quality of life and psychological condition
* About quality component:

A socio-demographic heel will be collected for each participant interviewed who has given no objection to participating in the study. His agreement on the recording of his voice will also collected.

For all participants, following data will be collected: Age, sex, occupation, date and duration of the interview, relationship with the Diapason 92 user (for family caregivers) and the recovery of socio-demographic data of the case report form (for users)

ELIGIBILITY:
Patient/Resident Inclusion Criteria

* Age ≥ 60 years old.
* (Group iso-resources) GIR ≤ 4
* Beneficiary of treatment by Diapason 92 or resident at EHPAD Aulagnier for more than 6 months.
* Not exhibiting severe disruptive behaviour disorders (on NPI-ES all FXG 12 and resonance 4 scores).
* Affiliate or entitled to a sickness insurance scheme
* Patient or legal representative expressed no objection

Patient/Resident Exclusion Criteria:

* Age < 60 years old
* GIR ˃ 4
* Not affiliated or entitled to a sickness insurance scheme
* Patient or legal representative did not express no objection

Professionals and caregivers Inclusion Criteria:

* Exercise within Diapason 92 device or be identified as assisting a Diapason 92 user or be a professional partner of Diapason 92 device
* Have expressed no objection to participating in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For quantitative component: we have two arms:
  * Diapason 92 arm: will be constitued by older patients with loss of autonomy, living at home and benefiting from Diapason 92 device
  * Control arm: will be constituted by people residing at the EHPAD (retirement home)
  For qualitative component: Study will cover 5 different populations since it concerns both:
  * Diapason 92 professionals who work directly with users
  * Daipason 92 Supervisory staff
  * Diapason 92 professional partners, including referring physicians.
  * The users
  * Non-professional helpers of users
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
Assessment of life quality according Nottingham Health Profile (NHP) scale | 12 months
  Difference in 12-month quality of life scores (Nottingham Health Profile) between the 2 groups (Diapason 92 and EHPAD).

SECONDARY OUTCOMES:
Assessment of the level of loss of autonomy of an elderly people according Autonomy, gerontology Iso Resources Group (AGGIR) scale | 12 months
Assessment of functional status according Lawton Instrumental Activities of Daily Living (IADL) Scale | 12 months
Assessment of activities of daily living, self-care, and independence according Activities of Daily Living (ADL) Scale | 12 months
Assessment of comorbidity according Charlson scale | 12 months
Assessment of cognitive function according Mini-Mental State Examination (MMSE) scale | 12 months
Assessment of disorders of disruptive behaviour according (NPI-ES) scale | 12 months
Assessment of geriatric depression according Geriatric Depression Scale (GDS) scale | 12 months
Measuring of burden of the close caregivers according Popular Caregiver Self-report measure Burden (ZARIT) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Phd Hanon, Principal Investigator — Geriatric department, Broca hospital (Paris)
Locations (1):
- Geriatric department , Broca Hospital, Paris, Île-de-France Region, France